CLINICAL TRIAL: NCT00511550
Title: Filgrastim-Mobilized Peripheral Blood Stem Cells for Allogeneic Transplantation With Unrelated Donors
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Other Study IDs: UC-2508; NCT00005930 (obsolete NCT alias)
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2007-07

CONDITIONS: Healthy
Keywords: peripheral blood stem cells; filgrastim-mobilized; allogeneic transplantation; Unrelated Donors for allogeneic transplantation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Peripheral blood stem cells (PBSCs) collected following stimulation with filgrastim are commonly used for autologous hematopoietic transplants. PBSCs are also now being used for some syngeneic and allogeneic hematopoietic transplants involving HLA-matched sibling donors. However, many issues remain unanswered about the use of PBSCs for allogeneic transplants and the effects of filgrastim on healthy individuals. The purpose of this study is to determine the effectiveness of filgrastim stimulated PBSCs in hematopoietic cell transplants involving unrelated donors and to determine the effects of this donation process on unrelated stem cell donors.

DETAILED DESCRIPTION:
This study establishes and evaluates a system to supply peripheral blood stem cell (PBSC)products for use in unrelated donor hematopoietic stem cell (HSC) transplantation. The protocol describes processes for donor identification, education and evaluation. Procedures for administration and monitoring of the stem cell mobilizing agent filgrastim are included. The study also describes procedures for the collection of PBSC products by leukapheresis and includes provisions for indefinite donor follow-up.

ELIGIBILITY:
Inclusion Criteria:

-Healthy adults

Exclusion Criteria:

* Pregnancy or uninterruptible breastfeeding.
* Sensitivity to filgrastim or to E. coli-derived recombinant protein products.
* History of autoimmune disorders, including rheumatic disease and thyroid disorders. Exception: As with bone marrow donations, donors with a history of thyroid disease who have undergone successful therapy may be suitable.
* History of deep vein thrombosis or pulmonary embolism.
* Thrombocytopenia <150 x 10(9)/L (<150,000/uL) at baseline evaluation.
* Current treatment with lithium. Drug interactions between filgrastim and lithium, which may potentiate the release of neutrophils, have not been full evaluated.
* Positive Hemoglobin-Solubility (e.g. SickleDex or equivalent) test.
* Donors receiving experimental therapy or investigational agents.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15
Dates: Start 2005-08; Study Completion 2007-11

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, M.D., Principal Investigator — University of California, San Francisco; John Miller, M.D.,Ph.D., Study Director — National Marrow Donor Program
Locations (1):
- University of California San Francisco Medical Center, San Francisco, California, United States